CLINICAL TRIAL: NCT04822779
Title: The Effectiveness of 4500 Joule Therapeutic Ultrasound in the Treatment of Calcific Tendinitis of the Shoulder
Brief Title: The Effectiveness of Therapeutic Ultrasound in the Treatment of Calcific Tendinitis of the Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Stjepan Čota, Stjepan Čota, MD, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHC Zagreb
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Rotator Cuff Tendinitis; Shoulder Pain; Musculoskeletal Diseases
Keywords: ultrasound therapy; rehabilitation; kinesiotherapy; diagnostic ultrasound
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: The research will be a double-blind randomized control prospective study.
Who Masked: Participant, Investigator
Masking Description: Randomization of patients will be performed before the intervention in the R software package and the results of the randomization will be known only to the therapist who will be involved in the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): This group will receive ultrasound therapy.
  Respondents will conduct individual medical-gymnastics: unloading pendular exercises if strength exercises cannot be started immediately, shoulder range exercises, and rotator cuff and scapula stabilizer exercises for 30 minutes per treatment.
  Interventions: Device: Sonopuls 490u, Enraf-Nonius, Rotterdam, Kingdom of the Netherlands
- Control Group (Sham Comparator): This group will receive sham ultrasound therapy.
  Respondents will conduct the same individual medical-gymnastics, as in the active group: unloading pendular exercises if strength exercises cannot be started immediately, shoulder range exercises, and rotator cuff and scapula stabilizer exercises for 30 minutes per treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Sonopuls 490u, Enraf-Nonius, Rotterdam, Kingdom of the Netherlands — Ultrasound therapy will be applied in continuous output, 1 MHz frequency, the intensity of 1.5 W / cm2, and duration 10 min per treatment, on the front of the shoulder, on the surface of 2 ultrasound heads (10 cm2).
  The position of the arm will be in adduction and internal rotation in RCT of the supraspinatus, adduction and external rotation of the arm in RCT of the subscapularis, and the position of the arm over the opposite shoulder in RCT of the infraspinatus.
  Arms: Active Group
Other: Placebo — Sham ultrasound therapy will be applied using a frequency of 0 Hz, intensity 0 W / cm2, 10 min per treatment.
  The position of the arm will be in adduction and internal rotation in RCT of the supraspinatus, adduction and external rotation of the arm in RCT of the subscapularis, and the position of the arm over the opposite shoulder in RCT of the infraspinatus.
  Arms: Control Group

SUMMARY:
Rotator cuff tendinitis (RCT) has a prevalence between 2.7 and 22%, and predominantly affects middle-aged women. The pathophysiology has not been fully elucidated to date. RCT is characterized by hydroxyapatite crystal deposition in the rotator cuff tendons. Approximately half of the patients with RCT have pain with acute or chronic shoulder mobility limitation. In some patients, RCT shows a tendency for spontaneous and rapid regression.

Diagnostic ultrasound (D-US) is a non-invasive, non-ionizing, and relatively inexpensive diagnostic imaging method that is safe and reliable in assessing rotator cuff pathology. It is very sensitive in the identification of calcifications that are shown in grayscale (B-mode) as hyperechoic structures with or without acoustic shadow. Based on ultrasound findings, Chiou HJ et al. have classified calcifications into 4 types: type I are arcuate, type II are fragmented or punctiform, type III are nodular, and type IV are cystic. Spontaneous resorption may occur with type III and IV calcifications. A positive Doppler signal (PD) surrounding the calcification is highly correlated with pain intensity.

According to the European Union of Medical Specialists-Physical and Rehabilitation Medicine (UEMS-PRM) guidelines, the basis of RCT therapy is individual medical gymnastics (IMG). It includes exercises aimed to restore full shoulder mobility, and improve rotator cuff and scapular stabilizer muscles strength. Other passive procedures are elective in the choice of treatment.

Ultrasound therapy is often used in the treatment of musculoskeletal shoulder pathology due to its thermal and non-thermal effects. It is considered that tissue heating stimulates healing (vasodilation, acceleration of the metabolism, and improvement of the viscoelastic properties of the connective tissue). The frequency of ultrasound therapy is selected depending on the desired depth of action (3 MHz for surface structures up to 2.5 cm depth, and 1 MHz for deeper structures, up to 5 cm depth). Pulse mode is commonly used in acute, while continuous in chronic conditions.

To date, only a few studies have evaluated the reduction in calcification size after ultrasound therapy. Although ultrasound therapy is routinely used in the treatment of painful shoulder, reviewing the results of research published so far, we can say that current knowledge about the effectiveness of ultrasound therapy in RCT is inconsistent (only several studies with a small number of subjects, different parameters of applied ultrasound therapy in terms of penetration depth, applied energy and duration of treatment). This indicates the need for further research.

DETAILED DESCRIPTION:
The research will be conducted in the Clinic for Rheumatic Diseases and Rehabilitation, University Hospital Center Zagreb. The research will be a double-blind randomized control prospective study. Randomization of patients will be performed before the intervention in the R software package and the results of the randomization will be known only to the therapist who will be involved in the treatment. The respondent and the examiner (doctor) will not be aware of in which group the patient is enrolled. All respondents will sign an informed consent before the study begins. Research has been approved by the Ethics Committee of Clinical Hospital Center Zagreb and the Ethics Committee of the School of Medicine, University of Zagreb.

The minimum sample size of a total of 42 subjects (21 in each group) was estimated according to the following characteristics: type 1 error (α = 0.05), power (1-β = 0.8) and effect size [(effect size) 0.2], with the expected use of two - way analysis of variance with two independent groups and two repeated measurements (2x2 ANOVA) with an estimated minimum correlation between repeated measurements r = 0.6.

Inclusion criteria are symptomatic RCT (VAS pain ≥ 4 + limited shoulder mobility) with D-US calcification size ≥ 5 mm, calcification type I and II according to Chiou HJ et al., and disease duration ≥ 2 months. Exclusion criteria are asymptomatic RCT or RCT with mild symptoms (VAS pain ≤ 3+ normal shoulder mobility), calcification size <5 mm, type III and IV calcification according to Chiou HJ et al., duration symptoms less than 2 months, rotator cuff tendon rupture, adhesive capsulitis, application of corticosteroids in the examined shoulder in the previous 3 months, glucocorticoid therapy, physical shoulder therapy in the previous 6 months, shock wave therapy in the previous 12 months, prior percutaneous calcification irrigation, current cervical or cervicobrachial pain syndrome, inflammatory rheumatic disease, scapular dyskinesia with positive assisted and repository scapular test, subacromial/subdeltoid bursitis, recent trauma or malignancy in malignant disease.

During the study, respondents will be able to relieve pain with paracetamol and/or tramadol. Respondents will keep a diary of analgesia, and nonsteroidal anti-inflammatory drugs (NSAIDs) and cryo massage will not be allowed due to their anti-inflammatory effect.

The investigators will record age, sex, dominant arm, height, body weight, body mass index, cigarette smoking, medications, physical activity (sports), and profession. Clinical examination will be performed on the first day and the last day of the therapy.

Ultrasound therapy (Sonopuls 490u, Enraf-Nonius, Rotterdam, Kingdom of the Netherlands) will be used with continuous output, frequency 1 MHz, intensity 1.5 W / cm2 and duration 10 min per treatment, on the front of the shoulder, on the surface of 2 ultrasound heads (10 cm2), with the position of the arm in adduction and internal rotation in RCT of the supraspinatus, adduction and external rotation of the arm in RCT of the subscapularis and the position of the arm over the opposite shoulder in RCT of the infraspinatus. Sham ultrasound therapy will be applied in the same way as ultrasound therapy, using a frequency of 0 Hz, intensity 0 W / cm2, 10 min per treatment. All respondents will conduct IMG that includes: unloading pendular exercises if strength exercises cannot be started immediately, shoulder range exercises, and rotator cuff and scapula stabilizer exercises for 30 minutes per treatment. The physiotherapist will apply ultrasound therapy and sham ultrasound therapy by slow circular motions through a neutral gel and perform IMG.

The respondent and the researcher will not know in which group the subject was randomized. The first group will receive ultrasound therapy and IMG, and the second sham ultrasound therapy and identical IMG for four weeks (5 therapies per week, a total of 20 therapies). The researcher will perform a standardized ultrasound examination of the shoulder of all respondents immediately before and immediately after the therapeutic intervention, measuring the size of the calcification. Another examiner will make an independent measurement of the calcification size. The final measure will take the average value of the two. The researcher will record a positive PD in the tendon around the calcification (on a scale of 0-3), assess the severity of shoulder pain at rest, at night and when moving using a visual analog scale of pain (VAS-pain; 0-10), measure passive and active shoulder mobility (goniometer in degrees), rotator cuff muscle strength (manual muscle test; 0-5), handgrip strength (hydraulic dynamometer in kg) and assess functional status using the Shoulder Pain and Disability Index (SPADI)). All respondents will be assessed the overall satisfaction of the therapeutic intervention using a five-point Likert scale.

The primary outcome of the study will be the change in calcification size measured by D-US before and after the intervention, while other outcome parameters are: reduction of pain, an increase of shoulder mobility, improvement of functional status, and overall satisfaction with rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic RCT (VAS pain ≥ 4 + limited shoulder mobility) with D-ultrasound calcification size ≥ 5 mm
* calcification type I and II according to Chiou HJ et al.
* disease duration ≥ 2 months

Exclusion Criteria:

* asymptomatic RCT or RCT with mild symptoms (VAS pain ≤ 3 + normal shoulder mobility)
* calcification size < 5 mm, type III and IV calcification according to Chiou HJ et al.
* duration symptoms less than 2 months
* rotator cuff tendon rupture
* adhesive capsulitis
* application of corticosteroids in the examined shoulder in the previous 3 months
* glucocorticoid therapy
* physical shoulder therapy in the previous 6 months
* shock wave therapy in the previous 12 months
* prior percutaneous calcification irrigation
* current cervical or cervicobrachial pain syndrome
* inflammatory rheumatic disease
* scapular dyskinesia with positive assisted and repository scapular test
* subacromial/subdeltoid bursitis
* recent trauma or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The change in calcification size measured by D-ultrasound before and after the intervention. | 4 weeks
  The researcher will perform an ultrasound examination of the shoulder immediately before and immediately after the therapeutic intervention. The size of the calcification will be measured according to the standard size measurement protocol, and another examiner will make an independent measurement. The final measure will take the average value of the two.

SECONDARY OUTCOMES:
To compare the effectiveness of therapeutic ultrasound in combination with individual medical gymnastics with the effectiveness of individual medical gymnastics in reducing pain. | 4 weeks
  The severity of shoulder pain will be assessed at rest, at night, and when moving using a visual analog scale of pain (VAS-pain; 0-10).
To compare the effectiveness of therapeutic ultrasound in combination with individual medical gymnastics with the effectiveness of individual medical gymnastics on increasing shoulder mobility. | 4 weeks
  Passive and active shoulder mobility will be measured with a goniometer.
To compare the effectiveness of therapeutic ultrasound in combination with individual medical gymnastics with the effectiveness of individual medical gymnastics on improving the functional status of the shoulder. | 4 weeks
  The functional status will be assessed using the Shoulder Pain and Disability Index (SPADI).
  SPADI consists of two dimensions, one for pain and the other for functional activities. The pain scale is summed up to a total of 50, while the disability scale is summed up to 80. The means of the two subscales are averaged to produce a total score ranging from 0 (the best) to 100 (the worst, more disability). The total SPADI score is expressed as a percentage.
To compare the effectiveness of therapeutic ultrasound in combination with individual medical gymnastics with the effectiveness of individual medical gymnastics on the overall satisfaction with the outcome of rehabilitation. | 4 weeks
  All respondents will be assessed the overall satisfaction of the therapeutic intervention using a five-point Likert scale (ranging from 1 to 5, 1 - completely dissatisfied, 2 - mostly dissatisfied, 3 - neither satisfied nor dissatisfied, 4 - mostly satisfied, 5 - fully satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- University Department for Rheumatology and Rehabilitation, Clinical Hospital Centre Zagre, Zagreb, City of Zagreb, Croatia

REFERENCES:
- [Background] Chiou HJ, Chou YH, Wu JJ, Hsu CC, Huang DY, Chang CY. Evaluation of calcific tendonitis of the rotator cuff: role of color Doppler ultrasonography. J Ultrasound Med. 2002 Mar;21(3):289-95; quiz 296-7. doi: 10.7863/jum.2002.21.3.289. PMID 11883540
- [Background] Varela E, Valero R, Kucukdeveci AA, Oral A, Ilieva E, Berteanu M, Christodoulou N; UEMS-PRM Section Professional Practice Committee. Shoulder pain management. The role of physical and rehabilitation medicine physicians. The European perspective based on the best evidence. A paper by the UEMS-PRM Section Professional Practice Committee. Eur J Phys Rehabil Med. 2013 Oct;49(5):743-51. PMID 24145232
- [Background] Alexander LD, Gilman DR, Brown DR, Brown JL, Houghton PE. Exposure to low amounts of ultrasound energy does not improve soft tissue shoulder pathology: a systematic review. Phys Ther. 2010 Jan;90(1):14-25. doi: 10.2522/ptj.20080272. Epub 2009 Nov 12. PMID 19910457
- [Background] Ebenbichler GR, Erdogmus CB, Resch KL, Funovics MA, Kainberger F, Barisani G, Aringer M, Nicolakis P, Wiesinger GF, Baghestanian M, Preisinger E, Fialka-Moser V. Ultrasound therapy for calcific tendinitis of the shoulder. N Engl J Med. 1999 May 20;340(20):1533-8. doi: 10.1056/NEJM199905203402002. PMID 10332014
- [Background] Williams JW Jr, Holleman DR Jr, Simel DL. Measuring shoulder function with the Shoulder Pain and Disability Index. J Rheumatol. 1995 Apr;22(4):727-32. PMID 7791172
- [Background] Philadelphia Panel. Philadelphia Panel evidence-based clinical practice guidelines on selected rehabilitation interventions for shoulder pain. Phys Ther. 2001 Oct;81(10):1719-30. PMID 11589645